CLINICAL TRIAL: NCT03768245
Title: Multi-Component School-Based Program On Obesity and Related Diseases, In A Multi-Ethnic Study
Brief Title: School-Based Program On Metabolic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, Paula Costa Urrutia, Ph.D, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 433.2016
Record Dates: First submitted 2018-12-04; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Cardiovascular Function; Kidney Diseases; Liver Diseases; Physical Fitness
Keywords: Body Mass Index; Glucose; Haemoglobin glycosylated; Blood Lipids; Liver Function; Kidney Function; Exercise; Physical activity
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Kidney Diseases; Liver Diseases; Motor Activity | interventions — Food Assistance

STUDY DESIGN:
Intervention Model Description: The intervention program is split into two groups of participants which receive two deferments treatments (Arms); treatment (Arm 1) is applied to all participants (n=800), while treatment 2 (Arm 2) is randomly applied just in the Mestizo group (n=117), i.e. schools and grade are randomly allocated in Arm 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behaviour (Experimental): Physical activity and the Health Education programs are applied.
  Interventions: Behavioral: Health Education and Physical activity program
- Nutrition (Active Comparator): In this Arm, the the Physical activity, the Health education and Nutrition program are applied.
  Interventions: Behavioral: Health Education and Physical activity program; Dietary Supplement: Nutrition Program

INTERVENTIONS:
Behavioral: Health Education and Physical activity program — Its objective is to empower children on healthy lifestyle, addressing four main topics: nutrition (i.e. healthy food, hydration), adequate quantities of food, physical activity, and self-monitoring. The program is implemented in the classroom through workshops planned and conducted by psychologists and nutritionists. A total of 12 workshops are planned, to be conducted once a week, and lasting 50 minutes each. The Physical activity program objective is to develop an active scholar environment, and consists of a moderate-vigorous activity, five days a week. The activities are divided into two types: (a) in the school backyard for 60 minutes, three times a week, and (b) in the classroom two days a week, for 15 minutes three times a day, adding up to 45 minutes daily.
Dietary Supplement: Nutrition Program — Its objective is to maintain lean mass, decrease fat mass and ensure mineral vitamins and fatty acids intake, maintain proper growth under National Specific Action Program: Food and Activity4. From total energy, a fat intake of 25-35%, carbohydrate intake of 45-65%, protein intake of 10-30%, and total calories are adjusted according to age. The Nutrition program consists of three meals: breakfast, a snack for a mid-morning playtime, and lunch at school. Food is prepared daily following sanitary and quality standards of Mexican official regulation. Breakfast is served 40 minutes before starting class time, lunch is served 40 minutes before leaving school.
  Arms: Nutrition

SUMMARY:
Mexico occupies the first place worldwide in childhood obesity. Its urban and indigenous communities present different levels of westernization which have triggered different epidemiological diseases. This study aims to treat and prevent obesity and related diseases. A school-based multi-component intervention program is developed in three ethnic groups with varying levels of westernization: Mestizos, Seris and Yaquis. Measurements are obtained to evaluate obesity, cardiovascular, diabetes risk, hepatic and renal function, and physical fitness. The intervention consists on Physical Activity (PA), Health Education (HE) and Nutrition (NP) programs carried out in six urban (Mestizo ethnic group) and indigenous schools (Seri and Yaqui ethnic groups). A total of 800 participants were part of the PA and HE programs (Education Arm), and 117 of them were also part of the NP program (Nutrition Arm). Measurement differences, after and before treatments are used to assess the intervention effect by age, sex, ethnicity, nutritional status, and treatments. Expanded access is not applicable to this study. The Government's Secretary of Education does not allow developing a plan to share individual data of participants.

DETAILED DESCRIPTION:
Participants from one preschool and 5 primary schools are included in the study. Participants are children between 5 and 12 years old from Sonora State, North of Mexico. Four urban schools of Mexican-Mestizos (from Hermosillo, capital city) and two indigenous schools, Seris (from Punta Chueca) and Yaquis (from Bahía de Lobos), participate in the program. Urban schools are randomly selected. Indigenous schools are hard to access, thus Seris and Yaquis school are chosen based on higher accessibility, and all grades from those schools (from first to sixth) are included. The intervention program consists of implementing Health Education, Nutrition and Physical Activity programs, and also parent involvement activities. All nutritionists, psychologists, and physical education teachers are prepared for their lessons during two weeks before the project implementation by the developers of the project (PCU and RA), who also supervise them. The intervention program is split into two Arms; the Education Arm, which is applied to all participants, and the Nutrition Arm, which includes the Health Education, the Physical Activity and also the Nutrition programs. The Nutrition program is randomly applied just in the Mestizo group, i.e. schools and grade are randomly allocated in Nutrition program. Anthropogenic and biochemical measurements are collected before (Measurements 1, M1) and after (Measurements 2, M2) treatments. Anthropogenic measurements are taken to all participants, while biochemical are randomly taken to 320 participants (includes all form Nutrition Arm). M1 and M2 are taken by the same team. Intervention effect is measured as the difference between M2 and M1, calculated as the difference (Dif) in M=M2-M1. Thus, negative DifM values indicate a decrease in the variable measured after the intervention, while positive DifM values indicate an increase in the variable. To assess the effect of age, sex, ethnic group (Mestizos, Seris, Yaquis), treatments (T1, T2) and nutritional status (Normal weight, Overweight+Obesity) in DifM (i.e. DifBMI), we perform Generalized Linear Models (GLMs) with Gaussian distribution(1). The initial model contains all single effects and all possible interactions of such explanatory variables. GLM simplification is done by stepwise deletion of the least significant terms. Subsequent models were generated by the stepwise removal of non-significant terms, and assessing each simplification with the Akaike information criterion (AIC) using the ΔAIC > 2 criterion(2). All models considered are subjected to the customary residual analyses and show a satisfactory fit (results not shown). All statistical analyses are carried out in R(3).

ELIGIBILITY:
Inclusion Criteria:

* Children from the selected grades and schools.
* Children who voluntarily accept participating in the program.
* Children whose parents must authorize their participation in the program, signing an informed consent document.

Exclusion Criteria:

• Participants with any incapacity to perform physical activity.

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Mean Change From Baseline In Body Mass Index At 12 Weeks | Up to 12 weeks
  Weight is measured kilograms using a Seca scale. Height is measured in meters cm using a standardized portable stadiometer Microtoise. Weight and height are be combined to report Body mass index (BMI) in kg/m^2. BMI cut-off points of normal weight, overweight and obesity are used as defined by World Health Organization5.
Mean Change From Baseline In Fasting Glucose Profile At 12 Weeks | Up to 12 weeks
  Blood samples are taken in the morning, after a 10-hours fasting to measure glucose in milligrams/decilitres.
Mean Change From Baseline In Fasting Glycated Haemoglobin At 12 Weeks | Up to 12 weeks
  Blood samples are taken in the morning, after a 10-hours fasting to glycated haemoglobin in percentage.
Mean Change From Baseline In Fasting Triglycerides At 12 Weeks | Up to 12 weeks
  Blood samples are taken in the morning, after a 10-hours fasting to triglycerides in milligrams/decilitres.
Mean Change From Baseline In Fasting Total Cholesterol At 12 Weeks | Up to 12 weeks
  Blood samples are taken in the morning, after a 10-hours fasting to total cholesterol in milligrams/decilitres.
Mean Change From Baseline In Fasting High Density Lipoprotein Cholesterol At 12 Weeks | Up to 12 weeks
  Blood samples are taken in the morning, after a 10-hours fasting to high density lipoprotein cholesterol in milligrams/decilitres.
Mean Change From Baseline In Fasting Low Density Lipoproteins Cholesterol At 12 Weeks | Up to 12 weeks
  Blood samples are taken in the morning, after a 10-hours fasting to low density lipoprotein cholesterol in milligrams/decilitres.
Mean Change From Baseline In Fasting Creatinine At 12 Weeks | Up to 12 weeks
  Description Blood samples were taken in the morning, after a 10-hours fasting to measure creatinine in milligrams/decilitres.
Mean Change From Baseline In Fasting Urea At 12 Weeks | Up to 12 weeks
  Description Blood samples were taken in the morning, after a 10-hours fasting to measure urea in milligrams/decilitres.
Mean Change From Baseline In Fasting Urea Nitrogen At 12 Weeks | Up to 12 weeks
  Blood samples were taken in the morning, after a 10-hours fasting to measure urea in milligrams/decilitres.
Mean Change From Baseline In Fasting Uric Acid At 12 Weeks | Up to 12 weeks
  Description Blood samples were taken in the morning, after a 10-hours fasting to measure uric acid in milligrams/decilitres.
Mean Change From Baseline In Fasting Glutamic Oxalacetic Transaminase At 12 Weeks. | Up to 12 weeks
  Blood samples were taken in the morning, after a 10-hour fast to measure glutamic oxalacetic transaminase measured in international units/litre (U/L).
Mean Change From Baseline In Fasting Glutamic Pyruvic Transaminase, At 12 Weeks | Up to 12 weeks
  Blood samples were taken in the morning, after a 10-hour fast to measure glutamic pyruvic transaminase measured in international units/litre (U/L).
Mean Change From Baseline In Fasting Bilirubin Profile, At 12 Weeks | Up to 12 weeks
  Blood samples were taken in the morning, after a 10-hour fast to measure direct, total and indirect bilirubin, measured in milligrams/decilitres.
Mean Change From Baseline In Indirect Of Maximum Oxygen Consumption At 12 Weeks | Up to 12 weeks
  The Course-Navette test are used to measure the indirect maximum oxygen consumption measured in milligrams/kilograms/minutes.
Mean Change From Baseline In Speed At 12 Weeks | Up to 12 weeks
  Speed is measured in meters/seconds using the 4x10 meters test.
Mean Change From Baseline In Strength-Resistance At 12 Weeks | Up to 12 weeks
  Strength-resistance is measured in number of repetition using the abdominal strength test, which consists of recording the maximum number of abdominals in 30 seconds.
Mean Change From Baseline In Power At 12 Weeks | Up to 12 weeks
  Power is measured in centimetres, using the long jump test which measures the explosive power of the lower body, and the vertical jump test, measured in centimetres, for measuring changes in leg power.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Costa-Urrutia, Ph.D, Study Director — Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Locations (1):
- Hospital Regional Adolfo Lopez Matelos, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costa-Urrutia P, Alvarez-Farina R, Abud C, Franco-Trecu V, Esparza-Romero J, Lopez-Morales CM, Rodriguez-Arellano ME, Valle Leal J, Colistro V, Granados J. Effect of multi-component school-based program on body mass index, cardiovascular and diabetes risks in a multi-ethnic study. BMC Pediatr. 2019 Nov 4;19(1):401. doi: 10.1186/s12887-019-1787-x. PMID 31679507
- See also: Describe the tests for physical fitness evaluation — https://sites.google.com/site/alphaprojectphysicalactivity